CLINICAL TRIAL: NCT01241214
Title: A Multi-center, Double-blind, Randomized, Placebo-controlled, Active Reference, Parallel-group, Study of ACT-129968 in Adult Patients With Seasonal Allergic Rhinitis
Brief Title: Study of ACT-129968 in Adult Patients With Seasonal Allergic Rhinitis
Acronym: SAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-060B202
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Seasonal allergic rhinitis; SAR; Allergic rhinitis; Allergies
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic; Hypersensitivity | interventions — 2-(2-(1-naphthoyl)-8-fluoro-3,4-dihydro-1H-pyrido(4,3-b)indol-5(2H)-yl)acetic acid; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Investigational drug - Dose 1 (Experimental)
  Interventions: Drug: ACT-129968
- Investigational drug - Dose 2 (Experimental)
  Interventions: Drug: ACT-129968
- Investigational drug - Dose 3 (Experimental)
  Interventions: Drug: ACT-129968
- Investigational Drug - Dose 4 (Experimental)
  Interventions: Drug: ACT-129968
- Active Matching Reference (Other)
  Interventions: Drug: Cetirizine
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: ACT-129968; Drug: Cetirizine; Drug: Placebo

INTERVENTIONS:
Drug: ACT-129968 — ACT-129968 (Dose 1, Dose 2, or Dose 3) or matching placebo administered orally twice daily
  Arms: Investigational drug - Dose 1; Investigational drug - Dose 2; Investigational drug - Dose 3; Matching Placebo
Drug: ACT-129968 — ACT-129968 (Dose 4) & matching placebo administered orally once daily
  Arms: Investigational Drug - Dose 4; Matching Placebo
Drug: Cetirizine — Ceterizine administered once daily
  Arms: Active Matching Reference; Matching Placebo
Drug: Placebo — Matching placebo administered twice daily.
  Arms: Matching Placebo

SUMMARY:
This study will assess the efficacy and safety of different doses of ACT-129968 in adult patients with seasonal allergic rhinitis, due to mountain cedar pollen.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 70 years.
* Clinical history of symptomatic seasonal allergic rhinitis associated with mountain cedar pollen for the last two years.
* Adequate exposure to mountain cedar pollen.
* Positive skin prick test to mountain cedar allergen within 12 months of screening.
* Sufficient nasal symptom score during a run-in period.

Exclusion Criteria:

* Non-allergic rhinitis.
* Bacterial or viral respiratory tract infection.
* Chronic respiratory disorders.
* Asthma requiring treatment other than inhaled short-acting Beta2-agonists.
* Ocular infections or surgery, nasal obstruction, nasal biopsy or surgery, sinus surgery or perforation.
* Smoking within the last year.
* Ongoing or recent treatment for seasonal allergic rhinitis.
* Initiation of allergen immunotherapy within 6 months of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To demonstrate a change in Daytime Nasal Symptom Score while taking Dose 3 of ACT-129968 versus placebo | Baseline to week 2

SECONDARY OUTCOMES:
To demonstrate a change in Daytime Nasal Symptom Score while taking either Dose 1, Dose 2, or Dose 4 of ACT-129968 verses placebo. | Baseline to week 2

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mangialaio, MD, Study Director — Actelion
Locations (7):
- United States (7):
  - Clinical Investigative Site 7905, Austin, Texas
  - Clinical Investigative Site 7907, Kerrville, Texas
  - Clinical Investigative Site 7903, New Braunfels, Texas
  - Clinical Investigative Site 7901, San Antonio, Texas
  - Clinical Investigative Site 7902, San Antonio, Texas
  - Clinical Investigative Site 7904, San Antonio, Texas
  - Clinical Investigative Site 7906, San Antonio, Texas

REFERENCES:
- [Derived] Ratner P, Andrews CP, Hampel FC, Martin B, Mohar DE, Bourrelly D, Danaietash P, Mangialaio S, Dingemanse J, Hmissi A, van Bavel J. Efficacy and safety of setipiprant in seasonal allergic rhinitis: results from Phase 2 and Phase 3 randomized, double-blind, placebo- and active-referenced studies. Allergy Asthma Clin Immunol. 2017 Apr 4;13:18. doi: 10.1186/s13223-017-0183-z. eCollection 2017. PMID 28392807